CLINICAL TRIAL: NCT04312178
Title: Combined Incentive Actions, Focusing on Primary Care, to Improve Cervical Cancer Screening in Women Residing in Socio-economically Disadvantaged and Untracked Geographical Areas: a Hybrid Efficacy and Implementation Trial
Acronym: RESISTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BARDOU DEPREV PREPS 2019
Record Dates: First submitted 2020-03-11; First posted 2020-03-18 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- return vaginal self-swab by mail (Other): Socially disadvantaged women who have received a vaginal self-swab and have to return it by mail
  Interventions: Other: no intervention
- financial incentive mail-back vaginal self-swab (Other): Socially disadvantaged women who have received a vaginal self-swab and have to return it by mail to obtain a cash incentive
  Interventions: Other: cash incentive
- handing over the vaginal swab to a professional (Other): Socially disadvantaged women who have received a vaginal self-swab and need to report it to a health professional
  Interventions: Other: no intervention; Other: return vaginal self-swab kit in person
- financial incentive the vaginal self-swab to a pro (Other): Socially disadvantaged women who have received a vaginal self-swab and have to report it to a health professional to obtain a cash incentive
  Interventions: Other: cash incentive; Other: return vaginal self-swab kit in person

INTERVENTIONS:
Other: cash incentive — cash incentive (20€ gift card)
  Arms: financial incentive mail-back vaginal self-swab; financial incentive the vaginal self-swab to a pro
Other: no intervention — no intervention
  Arms: handing over the vaginal swab to a professional; return vaginal self-swab by mail
Other: return vaginal self-swab kit in person — hand-delivered to a health care professional to encourage discussion of cervical cancer prevention
  Arms: financial incentive the vaginal self-swab to a pro; handing over the vaginal swab to a professional

SUMMARY:
Though potentially eradicable, cervical cancer is the 3rd most prevalent gynecological cancer, and the 2nd most prevalent before the age of 45. In France, approximately 1100 women die from cervical cancer each year, with 5-year survival strongly linked to the stage at diagnosis (93%, 63%, 35% and 16% for stages IA, IIA, IIIA and IVA). The prevention of cervical cancer is currently based on the combination of the vaccination of adolescent girls against the most common high-risk oncogenic human papilloma virus types and routine Papanicolaou cytology (Pap smears) every three years in women aged 25 to 65 years. The Health and Social Protection Survey conducted by the Institute for Research and Documentation in Health Economics in 2012 showed that young women who are not vaccinated have a socio-economic profile similar to that of women who do not attend cervical cancer screening, mainly: (i) the least screened women and least vaccinated young women live in low-income families; (ii) a low level of education is associated with fewer Pap smears; (iii) an absence of pap smears in mothers in the last three years is associated with less human papillomavirus vaccination in their daughters. Cervical cancer is the female cancer which, in France, has the highest proportion attributable to precariousness (21.1%), and for which there are strong territorial disparities in incidence.

Several factors may explain the difficulties in obtaining satisfactory rates of screening, such as geographical remoteness, the disengagement of general practitioners, economic constraints, or the geographical origin of women. Several countries such as the Netherlands have started routinely screening for cervical cancer by testing for human papillomavirus. This approach appears to be as beneficial as a screening campaign based on the Pap smear.

This approach has also just been validated by the French Health Authority which, in its public health recommendation dated 11 July 2019, states that "From the age of 30, the High Authority for Health recommends that the human papillomavirus test replace the cytological examination in primary screening for cervical cancer." In addition, this recommendation states that "Vaginal self-sampling is an alternative to cervical sampling by a health professional to detect the human papillomavirus test for undetected or under-detected women. This makes it easier to screen women who never get tested or who do not get tested as recommended." Moreover, the French Authority for Health specifies "In addition, complementary studies should be carried out to evaluate the feasibility and effectiveness of the different modalities for making these vaginal self-samples available, depending on the specific populations concerned (French Guyana, Mayotte, women living on the street, in shantytowns, migrant women, with limited access to health services, etc.)".

Two French trials show that when women ignored a letter sent to the home to invite them to receive a Pap smear, only 16 to 18% of women performed vaginal self-sampling when a kit was subsequently sent to their home. The delivery of a vaginal swab by a health professional does not increase adherence to screening compared to a reminder letter for a Pap smear (12% vs. 11.9%). Economic incentives may increase adherence to prevention policies, including those against human papillomavirus infections. They are often used to combat "present bias", i.e. the tendency to seek immediate, even limited, satisfaction rather than greater future satisfaction. A factorial design will be used to analyze the respective contribution of the delivery of the vaginal swab to a healthcare professional and an economic incentive of 20€. The hypothesis is that the the fact of returning the vaginal self-sampling to a health professional or an economic incentive will increase the participation of socially disadvantaged women in cervical cancer screening compared to simply returning it by mail without an incentive. It also postulate that health professionals will encourage women to perform a vaginal swab and adhere to the recommendations of the French Health Authority in case of a positive human papillomavirus test and that socially disadvantaged women will accept vaginal swabbing as a method of cervical cancer screening. Factors such as precariousness, life and migration paths, the socio-sanitary context, and the provision of primary care all play a role in prevention behaviors and may explain the heterogeneity of the observed effects.

ELIGIBILITY:
Inclusion Criteria:

* Woman between 30 and 65 years of age.
* Covered by a Regional Cancer Screening Coordination Centre for cervical cancer in 4 of the pilot departments for the implementation of this organised screening, and participating in the study.
* eligible for cervical cancer screening.
* Having not had a screening test for at least three years.
* Not having responded within 12 months to a letter inviting a screening test.
* Residing in a Block Grouped for Disadvantaged Statistical Information, quintiles 4 & 5 according to the European Deprivation Index classification.
* Covered by health insurance or AME

Exclusion Criteria:

* Ineligible for screening (e.g. hysterectomy or history of cervical cancer).
* Having returned a refusal coupon or NPAI (does not live at the address indicated)

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10446 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Proportion of women returning the HPV kit | 12 months after sending HPV kit
  Own effect of the economic incentive to get tested
Proportion of women visiting a health professional after receiving the kit and performing a pap smear or HPV test | 12 months after sending HPV kit
  The specific effect of encouraging women to get tested by a health Professional

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hassine A, Antoni G, Fender M, Slama K, Leandri FX, Fanon JL, Auvray C, Jaffar Bandjee MC, Traversier N, Fagour L, Rochaix L, Fiorina C, Pourette D, Opigez E, Dumont A, Bardou M, Study Group R. Combined incentive actions, focusing on primary care professionals, to improve cervical cancer screening in women living in socioeconomically disadvantaged geographical areas: a study protocol of a hybrid cluster randomised effectiveness and implementation trial- RESISTE. BMJ Open. 2022 Nov 23;12(11):e065952. doi: 10.1136/bmjopen-2022-065952. PMID 36418118